CLINICAL TRIAL: NCT03854162
Title: The Accuracy of Partially or Fully Guided Dental Implantation Performed With Dental Implantological Surgical Guide as Compared to Freehand Dental Implantation
Brief Title: A Study of a Surgical Guide for Dental Implantology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Szeged University (Other)
Collaborators: Alpha - Bio Tec Ltd. (Industry); dicomLAB Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IMP SMART 002
Record Dates: First submitted 2019-02-20; First posted 2019-02-26 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Dental Implantation, Endosseous; Dental Implants; Minimally Invasive Surgical Procedures; Surgery, Oral; Surgery, Computer-Assisted

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- FREEHAND (Active Comparator): For these cases, the regular protocol of the study site is observed. The operator has the plan at their disposal projected on a screen in the operating theater. The preparation of the bony bed and the insertion of the implant are performed freehand, without any guidance. The positions and directions are determined with the naked eye, observing the plan projected on the screen. At the end of the operation, the operation site is checked, hemostasis is provided, and the operator records the operation in the source documentation. 2±1 days later, a postoperative CT scan is taken. A follow-up visit is due 14±2 weeks later, after the osseointegration period.
  Interventions: Device: SMART Guide
- PILOT (Active Comparator): The SMART Guide surgical template is applied only in the initial phase of the operation. After having prepared soft tissue access, the template is placed, and only one drilling is performed through its sleeve, with the so-called pilot drill. The resulting borehole serves as directional guidance for the drills applied later in the process. Further drilling and implant insertion are both performed freehand. At the end of the operation, the operation site is checked, hemostasis is provided, and the operator records the operation in the source documentation. 2±1 days later, a postoperative CT scan is taken. A follow-up visit is due 14±2 weeks later, after the osseointegration period.
  Interventions: Device: SMART Guide
- PARTIAL GUIDE (Active Comparator): The only non-guided step is implant insertion, that is, all drilling happens through the SMART Guide surgical template. After having prepared soft tissue access, the guide is placed, and all drillings are performed through it, according to the surgical protocol. Here the depth of the bony bed is also determined, as the sleeve does not allow the drill to move any deeper than planned. At the end of the operation, the operation site is checked, hemostasis is provided, and the operator records the operation in the source documentation. 2±1 days later, a postoperative CT scan is taken. A follow-up visit is due 14±2 weeks later, after the osseointegration period.
  Interventions: Device: SMART Guide
- FULL GUIDE (Active Comparator): The SMART Guide surgical template is used for all steps of the operation, including the insertion of the implant. Apart from this, the procedure is exactly the same as described under "partial guide".
  Interventions: Device: SMART Guide

INTERVENTIONS:
Device: SMART Guide — The device manufactured according to a digital plan based on patient anatomy. Guiding sleeves are used, through which bone drills are applied. These sleeves sit in a plastic template that is a negative of the patient's dentition, so that the guide is properly stabilized during the operation. The position of the sleeves is calculated from the surgical plan in a way that they guide the drills in the planned position.The material of the template is medical plastic, the sleeves are made of medical steel.The device is applied by the dentist during the implant surgery. The template is placed on the remaining dentition of the patient and stabilized this way. By this, the sleeves are also stabilized in their planned position. Access through the soft tissue can be prepared through the given sleeve with a circular trephine, but the system also supports flap surgery. As access has been established, the dentist performs the surgical protocol as planned.

SUMMARY:
This is a prospective, adaptive, parallel study with four arms, which seeks to compare the accuracy of freehand and guided dental implantation surgeries. The basis of the comparison in each case is a digital plan, and that digital plan is compared to the actual postoperative status by computerized, three dimensional analysis.

DETAILED DESCRIPTION:
Osseointegration of endosseous implants has long been the focus of research in dental implantology, for obvious reasons. The use of Titanium became the standard quite soon, but it took decades of research to come up with the ideal shapes and surface modifications (both physical and chemical), so that today it is safe to assume that a properly placed commercially available dental implant will osseointegrate. The issue of osseointegration can thus be considered as practically resolved, and this traditional surface-oriented line of implant research now focuses on modifications to prevent complications, such as peri-implantitis (7). It must be seen, though, that for decades, the main goal was to keep the inserted implant in place, which pushed other important issues aside, such as the three- dimensional position of the inserted (and osseointegrated) implant in the bone. The lack of adequate imaging technologies also contributed to the paucity of research in this direction and clinicians - having no other option - started to plan implant positions in panoramic radiograms and perform implant surgeries relying on their ability to mentally merge those two- dimensional plans with patient anatomy. Today, this can be considered the standard approach to dental implant surgery.

The optimal positioning of the implant in the patient's bone is, in many respects, an issue of distinguished importance. First, the position of the implant has a profound impact on the fit of and stress distribution on the superstructure (i.e. crown or bridge), which, in turn, influences survival of the latter. The position of the implant also determines the distribution of stress in the supporting bone, which, ultimately, influences the long-term survival of the implant itself. In other words, a misplaced implant may be functional for some time, but will not survive in the long run. Finally, a misplaced implant can cause serious esthetic problems in the esthetic zone.

The rapid progress of information technology and digital image processing created a favorable environment for what may be called digital dentistry, including the computer-assisted, three- dimensional planning of implant surgery and the stereolithographic manufacturing of surgical guides based on such digital plans. Various systems and procedures exist, but cone-beam CT-based digital planning and the production of custom-made surgical guides are shared features. The studied SMART Guide guided system is unique in the sense that the entire process is digital, and no dental technical work is required.

The aim of such a guided system is to provide individualized patient care by a.) planning implant position(s) considering the individual patient anatomy and b.) manufacturing a custom-made surgical guide that serves to guide bone drills during the preparation of the bony bed of the planned implant. The custom-made guide is manufactured according to the digital plan. The result is a surgical accessory that exactly fits the remaining dentition of the patient (thereby stabilizing it) and ensures that the bony bed of the implant is prepared as planned. Meta-analyses show that these systems indeed allow highly accurate implant placement as compared to the plan. But is this any better than the traditional, freehand way of implant surgery and placement? Intuitively, one would answer yes, but, in fact, the question is quite difficult to answer, given the almost complete lack of studies on the accuracy of freehand implant placement. Therefore, one of the aims of this study is to make such a comparison. A further point is that in the everyday practice, surgical guides are used in either of the following three modalities: for the initiation of the bed preparation ("pilot"), for the initiation and the entire drilling process ("partial") and for the entire process including the insertion of the implant ("full"). It is assumed that the more extensively the guide is used, the more accurate the final implant position will be as compared to the plan. However, this is only an assumption, as no direct comparison is available. Therefore, it is also our aim to compare these modalities in terms of how accurate implantation they allow as compared to the plan.

The investigators hypothesize that all three guidance modalities will allow significantly more accurate implant placement than the freehand method. It is also hypothesized that the three modalities will differ in the accuracy they allow. In general, the investigators hypothesize that any form of guided implant surgery and placement yields significantly more accurate results than the freehand approach.

Primary aim Comparison of the accuracy of partially and fully guided implantation as indicated by angle deviation.

Secondary aims

The secondary aims of the study are as follows:

To compare the accuracy of the different methods as indicated by entry point deviation; To compare the accuracy of the different methods as indicated by apical deviation; To compare the accuracy of the different methods as indicated by volume overlap; To compare the influence of position (maxilla or mandible) on the accuracy of implantation; To assess the tolerability of implantation performed with surgical guide; To assess the safety of implantation performed with surgical guide; To assess dentist satisfaction with the surgical guide (custom questionnaire) To assess volunteer satisfaction (OHIP, custom questionnaire)

ELIGIBILITY:
Inclusion Criteria:

1. Male and female volunteers between 18 and 75 years of age
2. Partial edentulousness of the mandible or maxilla
3. Clinical situation fit for implantation as judged by the examining physician or principal investigator (satisfactory soft and hard tissue conditions and occlusion)
4. The volunteer communicates well with the examiner and compliance can be expected.

Informed consent.

Exclusion Criteria:

1. Pregnancy or lactation. Pregnancy is defined as the period beginning with conception and ending with birth.
2. Women in their childbearing age; by definition, any woman who - unless she uses effective contraception - can get pregnant in a physiological way. Eligibility for this study presupposes that the female subject will use effective contraception until 4 weeks after the end of her participation in the study. Effective contraception is defined as any of the following:

   * Barrier method: condom or diaphragm or cervical cap with spermicide. Note that spermicide in itself is not a barrier!
   * Full abstinence (if this is acceptable for the subject). Periodic abstinence, like the calendar- and temperature-based methods and interrupted intercourse are not acceptable.
   * Female sterilization: bilateral oophorectomy w/wo histerectomy or tubal ligation at least six weeks before participation in the study.
   * Sterilization of the male partner: vasectomy (no spermia in the ejaculate). The only partner of the participating female can be a male who has undergone vasectomy.
   * Hormonal contraception (oral, injection, or implanted); intrauterine device (IUD) or intrauterine system (IUS).
3. Any disease (including but not exclusively the diseases of metabolism, hematological diseases, diseases of the liver, the kidneys, the lungs, the nervous system, the endocrine organs, the heart and the intestines and infectious diseases) that, in the principal investigator's opinion, has a significant effect on the subject's general health and/or means an unacceptable risk factor for the person to receive implant treatment.
4. Known HIV, Hepatitis B or Hepatitis C infection.
5. Any internal or psychiatric disease that, in the opinion of the principal investigator, would risk compliance with the instructions or participation until the end of the study.
6. Participation in an experimental study or trial within four weeks before the randomization, or within five times the half-life of the experimental agent (whichever is longer)
7. Known allergy to any component of the implant or the implant guide
8. Limited mouth opening, which, in the examiner's opinion, would risk the success of the intervention
9. Increased gag reflex, poor tolerance of intraoral manipulation
10. Radiotherapy, irradiation of the mandible or the maxilla (either at the time of screening or in the past)
11. INR>2.5
12. Immunosuppressed state
13. Bisphosphonate treatment (either at the time of screening or in the past)
14. Alcohol or drug abuse
15. Habitual smoking
16. Untreated periodontitis
17. Retained root in the planned insertion site
18. Local infection
19. Lack of dental sanitation
20. Poor oral hygiene
21. Infection w/wo fever

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Angle deviation | 3 months
  The angle closed by the principal axis of the digitally implant as planned and the actual implant as placed expressed in degrees.

SECONDARY OUTCOMES:
Apical deviation | 3 months
  The deviation of the apical point of the placed implant from the apical point as planned in the three dimensional space, expressed in millimeters.
Hex deviation (also known as coronal deviation) | 3 months
  The angle closed by the principal axis of the digitally implant as planned and the actual implant as placed expressed in degrees (to one decimal).
Volume overlap | 3 months
  the overlap between the planned model implant and the placed implant as digitally Reconstructed from a postoperative cone-beam CT scan, expressed as a percentage.
Adverse events | 6 months
  The occurrence of adverse events, expressed as the number and seriousness of adverse events.
Volunteer satisfaction | 6 months
  The subjective satisfaction of volunteers as assessed by the Oral Health Impact Profile questionnaire, and a custom volunteer satisfaction questionnaire. Questionnaires administered three times during study period.
Dentist (operator) satisfaction | 3 months
  The subjective satisfaction of the operating dentist with the surgery as an experience, assessed by a custom questionnaire. Questionnaire administered after each surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Szeged, Department of Oral and Maxillofacial Surgery, Szeged, Hungary

REFERENCES:
- [Background] Smeets R, Stadlinger B, Schwarz F, Beck-Broichsitter B, Jung O, Precht C, Kloss F, Grobe A, Heiland M, Ebker T. Impact of Dental Implant Surface Modifications on Osseointegration. Biomed Res Int. 2016;2016:6285620. doi: 10.1155/2016/6285620. Epub 2016 Jul 11. PMID 27478833
- [Background] Yeo IS. Reality of dental implant surface modification: a short literature review. Open Biomed Eng J. 2014 Oct 31;8:114-9. doi: 10.2174/1874120701408010114. eCollection 2014. PMID 25400716
- [Background] Albrektsson T, Wennerberg A. Oral implant surfaces: Part 2--review focusing on clinical knowledge of different surfaces. Int J Prosthodont. 2004 Sep-Oct;17(5):544-64. PMID 15543911
- [Background] Albrektsson T, Wennerberg A. Oral implant surfaces: Part 1--review focusing on topographic and chemical properties of different surfaces and in vivo responses to them. Int J Prosthodont. 2004 Sep-Oct;17(5):536-43. PMID 15543910
- [Background] Mohammed Ibrahim M, Thulasingam C, Nasser KS, Balaji V, Rajakumar M, Rupkumar P. Evaluation of design parameters of dental implant shape, diameter and length on stress distribution: a finite element analysis. J Indian Prosthodont Soc. 2011 Sep;11(3):165-71. doi: 10.1007/s13191-011-0095-4. Epub 2011 Aug 20. PMID 22942576
- [Background] Ryu HS, Namgung C, Lee JH, Lim YJ. The influence of thread geometry on implant osseointegration under immediate loading: a literature review. J Adv Prosthodont. 2014 Dec;6(6):547-54. doi: 10.4047/jap.2014.6.6.547. Epub 2014 Dec 17. PMID 25551016
- [Background] Madi M, Zakaria O, Ichinose S, Kasugai S. Effect of Induced Periimplantitis on Dental Implants With and Without Ultrathin Hydroxyapatite Coating. Implant Dent. 2016 Feb;25(1):39-46. doi: 10.1097/ID.0000000000000331. PMID 26384099
- [Background] Gupta S, Patil N, Solanki J, Singh R, Laller S. Oral Implant Imaging: A Review. Malays J Med Sci. 2015 May-Jun;22(3):7-17. PMID 26715891
- [Background] Fayaz A, Geramy A, Memari Y, Rahmani Z. Effects of Length and Inclination of Implants on Terminal Abutment Teeth and Implants in Mandibular CL1 Removable Partial Denture Assessed by Three-Dimensional Finite Element Analysis. J Dent (Tehran). 2015 Oct;12(10):739-46. PMID 27252757
- [Background] Memari Y, Geramy A, Fayaz A, Rezvani Habib Abadi S, Mansouri Y. Influence of Implant Position on Stress Distribution in Implant-Assisted Distal Extension Removable Partial Dentures: A 3D Finite Element Analysis. J Dent (Tehran). 2014 Sep;11(5):523-30. Epub 2014 Sep 30. PMID 25628678
- [Background] Sagat G, Yalcin S, Gultekin BA, Mijiritsky E. Influence of arch shape and implant position on stress distribution around implants supporting fixed full-arch prosthesis in edentulous maxilla. Implant Dent. 2010 Dec;19(6):498-508. doi: 10.1097/ID.0b013e3181fa4267. PMID 21119354
- [Background] Behnaz E, Ramin M, Abbasi S, Pouya MA, Mahmood F. The effect of implant angulation and splinting on stress distribution in implant body and supporting bone: A finite element analysis. Eur J Dent. 2015 Jul-Sep;9(3):311-318. doi: 10.4103/1305-7456.163235. PMID 26430356
- [Background] Guerrero ME, Jacobs R, Loubele M, Schutyser F, Suetens P, van Steenberghe D. State-of-the-art on cone beam CT imaging for preoperative planning of implant placement. Clin Oral Investig. 2006 Mar;10(1):1-7. doi: 10.1007/s00784-005-0031-2. Epub 2006 Feb 16. PMID 16482455
- [Background] Menchini Fabris GB, Gelpi F, Giammarinaro E, Velasco Ortega E, Marconcini S, Covani U. A novel CAD/CAM-based surgical template for mandibular osteoplasty and guided implant insertion. J Biol Regul Homeost Agents. 2017 APR-JUN;31(2 Suppl. 2):99-106. PMID 28702970
- [Background] Bover-Ramos F, Vina-Almunia J, Cervera-Ballester J, Penarrocha-Diago M, Garcia-Mira B. Accuracy of Implant Placement with Computer-Guided Surgery: A Systematic Review and Meta-Analysis Comparing Cadaver, Clinical, and In Vitro Studies. Int J Oral Maxillofac Implants. 2018 January/February;33(1):101-115. doi: 10.11607/jomi.5556. Epub 2017 Jun 20. PMID 28632253
- [Background] Tahmaseb A, Wismeijer D, Coucke W, Derksen W. Computer technology applications in surgical implant dentistry: a systematic review. Int J Oral Maxillofac Implants. 2014;29 Suppl:25-42. doi: 10.11607/jomi.2014suppl.g1.2. PMID 24660188